CLINICAL TRIAL: NCT05451888
Title: Assessing Effects of Mineral-rich Floatation Spa Treatment on Mood and Psychological Health Outcomes
Acronym: USS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Daniel Lamport, Associate Professor Daniel Lamport, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UReading Spa Study
Record Dates: First submitted 2022-06-16; First posted 2022-07-11 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Mood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Celestial Floatation Pool (Experimental)
  Interventions: Behavioral: Spa treatment
- Dead Sea Salt Pool (Experimental)
  Interventions: Behavioral: Spa treatment
- Balneotherapy Control Pool (Active Comparator)
  Interventions: Behavioral: Spa treatment

INTERVENTIONS:
Behavioral: Spa treatment — A 40 minute period of lying in the spa treatment pool

SUMMARY:
This is a randomised parallel groups trial in healthy human adults exploring whether 8 weeks of treatment in various different spa pools is associated with benefits for mood and other psychological outcomes. Outcome measures will be taken at the beginning and the end of the 8 week period. In addition, outcome measures will be taken after the first spa session to assess acute effects.

DETAILED DESCRIPTION:
This experiment is investigating whether mineral-rich floatation spa treatments influence mood and psychological health outcomes. The study will be undertaken at Nirvana Spa in Wokingham over a duration of 8 weeks for each participant. Participants will be randomly allocated to one of three experimental groups. Each group will be assigned to a different mineral-rich spa treatment pool; either a Celestial Floatation pool, Dead Sea Salt Therapy pool, or a control pool which does not contain any minerals (Balneotherapy pool). Participants will undergo one 40-minute treatment, once a week for 8 weeks. The recommended duration for Dead Sea Salt and Celestial floatation pool sessions are 30-40 minutes, thus this study will reflect everyday consumer behaviour. A follow-up assessment of the outcome measures will take place 2 weeks after cessation of treatment to assess possible carry-over effects.

Specifically, there are four research aims of the study;

1. To investigate the effects of regular weekly treatment in the Celestial Floatation Pool on mood outcomes including positive and negative affect, anxiety, depression, and stress.
2. To investigate the effects of regular weekly treatment in the Dead Sea Salt Therapy pool on mood outcomes including positive and negative affect, anxiety, depression, and stress.
3. To investigate the effects of a single 40-minute treatment in the Celestial Floatation Pool and the Dead Sea Salt Therapy pool on mood outcomes including positive and negative affect, anxiety and stress.
4. Do any beneficial effects of spa treatment persist beyond cessation of treatment?

Outcome measures will be used to assess mood and psychological health outcomes both at the beginning (baseline) and at the end (8 weeks) of each treatment (see procedures). In addition, outcome measures will be taken immediately after the first spa treatment to assess acute effects. Specifically, the outcome measures are:

* Positive and Negative Affect using the PANAS-X. This will be a well-established measure of how positive and negative an individual is feeling (these are two separate outcome measures).
* Subjective mood with the Immediate Mood Scaler. This is a recently published novel 22-item measure developed to assess dynamic components of mood. Participants rate their current mood state on a continuum using 7-point Likert scales (eg, happy-sad, distracted-focused, sleepy-alert, fearful-fearless. For each item, an integer score between 1 and 7 is derived. The total score for this scale is the sum of the scores on all 22 items.
* Stress using the Perceived Stress Scale.
* Anxiety with the GAD-7 and the Spielberger State Anxiety Inventory.
* Depression with the PHQ-8
* Sleep quality with the Pittsburgh Sleep Quality Index (PSQI)
* Experience of spa use will be captured using qualitative and quantitative questions on their enjoyment of the spa intervention and ease of use.

ELIGIBILITY:
Inclusion Criteria:

Any adult

Exclusion Criteria:

Any diagnosed mental health conditions or physical conditions/injuries (including those still undergoing physiotherapy for a previous condition or injury), arthritis and previous regular use of spa treatments which is defined as use of spa facilities once a month or more over the previous 8 weeks. The rational for these exclusion criteria is that the spa is known to benefit injury and joint pain recovery. This is not a mechanism of interest for this study, therefore we want to exclude these participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Positive Affect (chronic) | Change between baseline and 8 weeks
  This will be a well-established measure of how positive an individual is feeling measured using the PANAS-X questionnaire
Negative Affect (chronic) | Change between Baseline and 8 weeks
  This will be a well-established measure of how negative an individual is feeling measured using the PANAS-X questionnaire

SECONDARY OUTCOMES:
Subjective mood | Change between baseline and 8 weeks
  Assessed with the Immediate Mood Scaler
Subjective Stress | Change between baseline and 8 weeks
  Assessed with the Perceived Stress Scale
Anxiety | Change between baseline and 8 weeks
  Assessed with the GAD-7 and the Spielberger State Anxiety Inventory
Depression | Change between baseline and 8 weeks
  PHQ-8
Sleep Quality | Change between Baseline and 8 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Subjective experience of the spa | At 8 weeks
  captured using qualitative and quantitative questions on their enjoyment of the spa intervention and ease of use.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided